CLINICAL TRIAL: NCT05446103
Title: The Acute Effect of Upper Limb Low Load Blood Flow Restriction Training (BFRT) on Hypoalgesia. A Randomized Controlled Trial
Brief Title: The Hypoalgesic Effects of Low Load Blood Flow Restriction Training (BFRT)
Acronym: BFRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Stefanos Karanasios, Principal Investigator, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SK1
Record Dates: First submitted 2022-06-28; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: blood flow restriction; pressure pain threshold; exercise; training
MeSH Terms: conditions — Motor Activity | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Using sham blood flow restriction (A cuff will be placed on the arm with minimum pressure <20% of arterial occlusive pressure)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR (Experimental): 20 healthy individuals will be assigned to perform elbow flexion exercises with low-load resistance BFR training (30% of 1 RM)
  Interventions: Other: Blood flow restriction training
- Sham BFR (Sham Comparator): 20 healthy individuals will be assigned to perform elbow flexion exercises with high-load resistance training with sham BFR (65% of 1 RM)
  Interventions: Other: Sham Blood flow restriction training

INTERVENTIONS:
Other: Blood flow restriction training — After warming up, the load is set at 80% of the predicted 1Repetition Maximum (RM) for elbow flexors. Following each successful repetition, the load is increased by 0.5 to 1kg until patients: fail to execute the exercise through the entire range of motion; used improper form to complete the repetition; needed assistance; reported pain. We will allow a 2-3 min of rest between each attempt to ensure recovery.
  The session starts by calculating the arterial occlusion pressure in the standard anatomical position. Participants rest in the standing position for 3-5 minutes before measurement to ensure restoration of blood flow circulation and a cuff is placed in the most proximal part of their dominant upper-limb. BFR application is conducted by using an automatic personalized tourniquet system (Mad-Up Pro, France). An 40% occlusion pressure is set and subjects perform 4 sets of elbow flexion (30-15-15-15 reps) using 30% of 1 RM
  Arms: BFR
Other: Sham Blood flow restriction training — After warming up, the load is set at 80% of the predicted 1Repetition Maximum (RM) for elbow flexors. Following each successful repetition, the load is increased by 0.5 to 1kg until patients: fail to execute the exercise through the entire range of motion; used improper form to complete the repetition; needed assistance; reported pain. We will allow a 2-3 min of rest between each attempt to ensure recovery.
  The session starts by calculating the arterial occlusion pressure in the standard anatomical position. Participants rest in the standing position for 3-5 minutes before measurement to ensure restoration of blood flow circulation and a cuff is placed in the most proximal part of their dominant upper-limb. BFR application is conducted by using an automatic personalized tourniquet system (Mad-Up Pro, France). An <20% of occlusion pressure is set and subjects perform 4 sets of 10 reps of elbow flexion using 65% of 1 RM
  Arms: Sham BFR

SUMMARY:
A randomized controlled trial comparing the immediate effects of upper limb low-load blood flow restriction training (BFRT) with high load sham-BFRT on hypoalgesia and perceptual response in healthy adults

DETAILED DESCRIPTION:
Healthy individuals will be randomized to one of two groups. A target of 40 patients for enrollment has been set for 80% power, p<0.05 (Effect size= 1). A single Intervention will be used (40 minutes).

Intervention Group: A single exercise of elbow flexion with Blood Flow Restriction (30-15-15-15 reps) using 30% of 1 Repetition Maximum.

Control Group: A single exercise of elbow flexion with sham Blood Flow Restriction (4x10 reps) using 65% of 1 Repetition Maximum.

Primary outcome: pressure pain thresholds on quadriceps, biceps, lateral epicondyle and upper trapezius (bilateral).

Secondary outcomes: difference in perceptual response (exertion), change in blood pressure

ELIGIBILITY:
Inclusion Criteria:

* BMI< 30
* able to perform full elbow flexion and extension

Exclusion Criteria:

* shoulder tendinopathy,
* cervical radiculopathy,
* rheumatoid arthritis,
* neurological deficit,
* serious cardiovascular diseases,
* venous deficiency,
* history of heart surgery,
* cancer history,
* breast surgery,
* orthopaedic surgeries during the last 6 months,
* thrombosis,
* diabetes,
* body mass Index ≥ 30,
* Crohn syndrome,
* family or personal history of pulmonary embolism

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold | Baseline and 30 minutes
  Changes between pre- and post- intervention in Pressure Pain Threshold will be measured using bilateral sites on quadriceps, upper trapezius, lateral epicondyle and biceps. The COMPACT DIGITAL ALGOMETER CAPACITIES TO: 100 lbf / 50 kgf / 500 N, will be used by an independent assessor. The assessor will be blinded to participants' group.

SECONDARY OUTCOMES:
Rating of perceived exertion | At the end of the 1st, 2nd, 3rd and 4th set ( after 1, 2, 3 and 4 minutes respectively)
  Changes between each set of exercise of Perceived Exertion. Measurements will include a Borg 6-20 scale based on the strain and fatigue in muscles. 6 means 'no exertion at all' and 20 means 'maximal
Blood pressure | Baseline and 30 minutes
  Changes in systolic and diastolic blood pressure between pre and post intervention. Blood pressure will be measured in a seated position using a electronic device (Omron)

CONTACTS AND LOCATIONS:
Overall Officials: George Gioftsos, PhD, Study Chair — University of West Attica; Stefanos Karanasios, PhD, Study Director — University of West Attica; Alexia Sozeri, MSc, Principal Investigator — University of West Attica
Locations (1):
- University of West Attica, Aigáleo, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bowman EN, Elshaar R, Milligan H, Jue G, Mohr K, Brown P, Watanabe DM, Limpisvasti O. Upper-extremity blood flow restriction: the proximal, distal, and contralateral effects-a randomized controlled trial. J Shoulder Elbow Surg. 2020 Jun;29(6):1267-1274. doi: 10.1016/j.jse.2020.02.003. PMID 32423577
- [Background] Gearhart RE, Goss FL, Lagally KM, Jakicic JM, Gallagher J, Robertson RJ. Standardized scaling procedures for rating perceived exertion during resistance exercise. J Strength Cond Res. 2001 Aug;15(3):320-5. PMID 11710658
- [Background] Hughes L, Patterson SD. The effect of blood flow restriction exercise on exercise-induced hypoalgesia and endogenous opioid and endocannabinoid mechanisms of pain modulation. J Appl Physiol (1985). 2020 Apr 1;128(4):914-924. doi: 10.1152/japplphysiol.00768.2019. Epub 2020 Feb 27. PMID 32105522
- [Background] Hughes L, Patterson SD, Haddad F, Rosenblatt B, Gissane C, McCarthy D, Clarke T, Ferris G, Dawes J, Paton B. Examination of the comfort and pain experienced with blood flow restriction training during post-surgery rehabilitation of anterior cruciate ligament reconstruction patients: A UK National Health Service trial. Phys Ther Sport. 2019 Sep;39:90-98. doi: 10.1016/j.ptsp.2019.06.014. Epub 2019 Jul 2. PMID 31288213
- [Background] Korakakis V, Whiteley R, Epameinontidis K. Blood Flow Restriction induces hypoalgesia in recreationally active adult male anterior knee pain patients allowing therapeutic exercise loading. Phys Ther Sport. 2018 Jul;32:235-243. doi: 10.1016/j.ptsp.2018.05.021. Epub 2018 May 31. PMID 29879638
- [Background] Korakakis V, Whiteley R, Giakas G. Low load resistance training with blood flow restriction decreases anterior knee pain more than resistance training alone. A pilot randomised controlled trial. Phys Ther Sport. 2018 Nov;34:121-128. doi: 10.1016/j.ptsp.2018.09.007. Epub 2018 Sep 19. PMID 30268966
- [Background] Lacruz ME, Kluttig A, Kuss O, Tiller D, Medenwald D, Nuding S, Greiser KH, Frantz S, Haerting J. Short-term blood pressure variability - variation between arm side, body position and successive measurements: a population-based cohort study. BMC Cardiovasc Disord. 2017 Jan 18;17(1):31. doi: 10.1186/s12872-017-0468-7. PMID 28100183
- [Background] Calvo Lobo C, Romero Morales C, Rodriguez Sanz D, Sanz Corbalan I, Sanchez Romero EA, Fernandez Carnero J, Lopez Lopez D. Comparison of hand grip strength and upper limb pressure pain threshold between older adults with or without non-specific shoulder pain. PeerJ. 2017 Feb 9;5:e2995. doi: 10.7717/peerj.2995. eCollection 2017. PMID 28289561
- [Background] Minniti MC, Statkevich AP, Kelly RL, Rigsby VP, Exline MM, Rhon DI, Clewley D. The Safety of Blood Flow Restriction Training as a Therapeutic Intervention for Patients With Musculoskeletal Disorders: A Systematic Review. Am J Sports Med. 2020 Jun;48(7):1773-1785. doi: 10.1177/0363546519882652. Epub 2019 Nov 11. PMID 31710505
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448